CLINICAL TRIAL: NCT05524285
Title: Safety Study of Intracranial Support Catheter and Guide Catheter for Stent-Assisted Embolization in the Treatment of Intracranial Aneurysms: A Prospective, Multicenter, Randomized, Open, Controlled, Superiority Trial
Brief Title: Safety Study of Intracranial Support Catheter and Guide Catheter for Stent-Assisted Embolization in the Treatment of Intracranial Aneurysms
Acronym: SAFETI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 2022-0505
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-08

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intracranial Support Catheter
  Interventions: Device: Intracranial Support Catheter
- control group (Active Comparator): Guide Catheter
  Interventions: Device: Guide Catheter

INTERVENTIONS:
Device: Intracranial Support Catheter — Endovascular procedure using the intracranial support catheter which approved by NMPA
  Arms: experimental group
Device: Guide Catheter — Endovascular procedure using the guide catheter which approved by NMPA
  Arms: control group

SUMMARY:
The purpose of this study is to evaluate the safety differences between intracranial support catheter and guide catheter for stent-assisted embolization in the treatment of unruptured intracranial aneurysms in the anterior circulation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open, controlled, superiority trial carried out in 9 research centers over China. Patients are randomized 1:1 to therapy either intracranial support catheter or guide catheter. Taking the guide catheter as a control, to evaluate whether the safety of intracranial support catheter for stent-assisted embolization in the treatment of unruptured intracranial aneurysms in the anterior circulation is superior than that of the control.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 and≤70 years, any gender;
* Preoperative modified Rankin Scale (mRS) score 0-2;
* Subject has an unruptured intracranial aneurysm in the anterior circulation diagnosed by DSA/CTA/MRA (accept the results from other hospital)；
* No intracranial hemorrhage and recent cerebral infarction (DWI indicates hyperintense lesions) are founded by preoperative MRI+DWI;
* Subject is assessed as suitable for stent-assisted coil embolization (SACE) treatment (except flow diverter stent);
* Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form.

Exclusion Criteria:

* Inadequate antiplatelet therapy before surgery (more than 3 days);
* Subject with atrial fibrillation, patent foramen ovale, atrial septal defect, ventricular septal defect, and other diseases causing cardiogenic embolism;
* Inability to perform cranial MRI+DWI preoperatively and within 48 hours postoperatively;
* Hypertension that does not respond well to medical treatment (systolic blood pressure>185 mmHg and/or diastolic blood pressure>110 mmHg);
* Preoperative active bleeding or bleeding tendency (INR>3);
* Random blood glucose<2.7mmol/L or >22.2mmol/L;
* Heart, lung, liver and kidney failure or other serious diseases (intracranial tumor, intracranial arteriovenous malformation, severe infection, DIC, previous myocardial infarction, history of severe psychosis, etc.);
* Subject who will not cooperate or tolerate interventional operation;
* Anticipated life expectancy<1 year;
* Allergy, resistance or contraindication to one or more of the following: contrast agents, anesthetics, antiplatelet drugs, anticoagulants;
* Participated or participating in another drug or device clinical trial within 1 month prior to enrollment;
* Pregnant or breast-feeding woman;
* Other circumstances judged by researchers that are not suitable for enrollment;
* Catheter could not pass through due to obvious intracranial vessel stenosis or tortuosity determined from imaging;
* Multiple aneurysms and more than one aneurysm requiring treatment;
* The aneurysm body has arterial branches.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic cerebral infarction within 48 hours postoperation | within 48 hours postoperation
  Symptomatic cerebral infarction is defined as NIHSS score increased by≥4 points compared with preoperation, along with imaging confirmed to be caused by infarction.

SECONDARY OUTCOMES:
Incidence of new-onset DWI positive postoperation | within 48 hours postoperation
  New-onset DWI positive is defined as any new hyperintense lesions.
Rate of catheter-related complications | Intraoperation
  Catheter-related complications are defined as vasospasm, vascular dissection, etc. which caused by catheter during operation.
Incidence of symptomatic cerebral infarction at 7 days postoperation or at discharge | 7 days postoperation or discharged
  Symptomatic cerebral infarction is defined as NIHSS score increased by≥4 points compared with preoperation, along with imaging confirmed to be caused by infarction.
Rate of mRS score 0-2 at 90 days | 90±14 days postoperation
  mRS score 0-2 indicates good prognosis.
All-cause mortality within 90 days | up to 90 days
  All-cause mortality is defined as all deaths due to any cause.
Incidence of Adverse Events (AE) | up to 90 days
Incidence of Serious Adverse Events (SAE) | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (9):
- China (9):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang